CLINICAL TRIAL: NCT05870696
Title: Evaluation of the Serum Metabolite Based PrecogColo Dx Test for Advanced Colorectal Neoplasia Screening
Brief Title: the Serum Metabolite Based PrecogColo Dx Test for Advanced Colorectal Neoplasia Screening
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PekingUTH-ding36
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Adenoma
Keywords: colorectal adenomas; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- negative: normal:no findings on colonoscopy hyperplastic polyps: inflammatory or hyperplastic polyps low-risk adenoma:1 or 2 adenoma(s), ≤10 mm in size, non-advanced
  Interventions: Diagnostic Test: PrecogColo Dx test
- Positive: advanced adenoma Advance adenoma, including the following subcategories:
  * Adenoma with carcinoma in situ/high grade dysplasia, any size
  * Adenoma, villous growth pattern (>25%), any size
  * Adenoma > 1.0 cm in size
  * Serrated lesion, > 1.0 cm in size early stage CRC: CRC stage I advanced stage CRC: CRC stage II-IV
  Interventions: Diagnostic Test: PrecogColo Dx test

INTERVENTIONS:
Diagnostic Test: PrecogColo Dx test — the serum metabolite based PrecogColo Dx test for advanced colorectal neoplasia Screening, including advanced adenoma and colorectal cancer

SUMMARY:
This study is to Evaluate the diagnostic sensitivity of the serum metabolite based PrecogColo Dx test for advanced colorectal neoplasia Screening, including advanced adenoma and colorectal cancer. There are two steps in this study. Firstly, the diagnostic model is established based on tumor-specific and gut-microbiome related serum metabolites. Secondly, the sensitivity, specificity and accuracy of the diagnostic model is evaluated in detecting advanced adenoma and colorectal cancer stages in an independent multi-centered cohort.

DETAILED DESCRIPTION:
Subjects aged >45 at average risk for development of CRC will be enrolled. Subjects will complete the PrecogColo Dx test, followed by completion of a screening colonoscopy. . Results from PrecogColo Dx test were compared to the results of an optical colonoscopic examination, and histopathological diagnosis of all significant lesions discovered during the colonoscopy, in order to determine the sensitivity for CRC and advanced adenoma, respectively, as well as determining specificity of non-advanced neoplasia individuals. Histopathological results from biopsied tissue or excised lesions were categorized based on the most clinically significant lesion present by a central pathologist.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 45 years of age at the time of enrollment.
2. Subject presents for a screening colonoscopy.
3. Subject has no symptoms or signs that require immediate, or near term, referral for diagnostic or therapeutic colonoscopy.
4. Subject is able and willing to sign informed consent.

Exclusion Criteria:

1. Patients received tumor treatment prior to the drawn of blood sample, including surgical resection, neoadjuvant chemotherapy, neoadjuvant chemoradiotherapy and targeted therapy.
2. Patients received antibiotics within 2 weeks.
3. Patients with indications of emergency surgery, including bleeding, obstruction and perforation.
4. Patients who are positive for Human Immunodeficiency Virus (HIV).
5. Patients with abnormal liver and kidney function.
6. Patients with the history of inflammatory bowel disease.
7. Patients who had history of other malignancies.
8. Subject has a diagnosis or medical history of any of the following conditions:

   1. Familial adenomatous polyposis (also referred to as "FAP", including attenuated FAP and Gardner's syndrome)
   2. Hereditary non-polyposis CRC syndrome (also referred to as "HNPCC" or "Lynch Syndrome")

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 45 years of age and older who are eligible for colorectal cancer screening and scheduled for a screening colonoscopy. Approximately 2,000 subjects will be targeted for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2024-02-27 (Estimated); Study Completion 2024-02-27 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Evaluations | 2 weeks
  Lower bound of the 95% one-sided confidence interval of PrecogColo Dx Sensitivity for CRC was greater than 65%, and lower bound of the 95% one-sided confidence interval of PrecogColo Dx specificity for non-advanced neoplasia (including normal, non-adenomas polyps and low risk adenoma) was greater than 85%.

CONTACTS AND LOCATIONS:
Overall Officials: shigang ding, doctor, Principal Investigator — Peking University Third Hospital
Locations (6):
- China (6):
  - Beijing Huaxin Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Aerospace Center Hospital, Beijing, Beijing Municipality
  - Beijing haidian hospital, Beijing, Beijing Municipality
  - Peking university third hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Vatandoost N, Ghanbari J, Mojaver M, Avan A, Ghayour-Mobarhan M, Nedaeinia R, Salehi R. Early detection of colorectal cancer: from conventional methods to novel biomarkers. J Cancer Res Clin Oncol. 2016 Feb;142(2):341-51. doi: 10.1007/s00432-015-1928-z. Epub 2015 Feb 17. PMID 25687380
- [Background] Doubeni CA, Corley DA, Quinn VP, Jensen CD, Zauber AG, Goodman M, Johnson JR, Mehta SJ, Becerra TA, Zhao WK, Schottinger J, Doria-Rose VP, Levin TR, Weiss NS, Fletcher RH. Effectiveness of screening colonoscopy in reducing the risk of death from right and left colon cancer: a large community-based study. Gut. 2018 Feb;67(2):291-298. doi: 10.1136/gutjnl-2016-312712. Epub 2016 Oct 12. PMID 27733426
- [Background] Niedermaier T, Balavarca Y, Brenner H. Stage-Specific Sensitivity of Fecal Immunochemical Tests for Detecting Colorectal Cancer: Systematic Review and Meta-Analysis. Am J Gastroenterol. 2020 Jan;115(1):56-69. doi: 10.14309/ajg.0000000000000465. PMID 31850933
- [Background] Janney A, Powrie F, Mann EH. Host-microbiota maladaptation in colorectal cancer. Nature. 2020 Sep;585(7826):509-517. doi: 10.1038/s41586-020-2729-3. Epub 2020 Sep 23. PMID 32968260
- [Background] Yachida S, Mizutani S, Shiroma H, Shiba S, Nakajima T, Sakamoto T, Watanabe H, Masuda K, Nishimoto Y, Kubo M, Hosoda F, Rokutan H, Matsumoto M, Takamaru H, Yamada M, Matsuda T, Iwasaki M, Yamaji T, Yachida T, Soga T, Kurokawa K, Toyoda A, Ogura Y, Hayashi T, Hatakeyama M, Nakagama H, Saito Y, Fukuda S, Shibata T, Yamada T. Metagenomic and metabolomic analyses reveal distinct stage-specific phenotypes of the gut microbiota in colorectal cancer. Nat Med. 2019 Jun;25(6):968-976. doi: 10.1038/s41591-019-0458-7. Epub 2019 Jun 6. PMID 31171880
- [Background] Chen F, Dai X, Zhou CC, Li KX, Zhang YJ, Lou XY, Zhu YM, Sun YL, Peng BX, Cui W. Integrated analysis of the faecal metagenome and serum metabolome reveals the role of gut microbiome-associated metabolites in the detection of colorectal cancer and adenoma. Gut. 2022 Jul;71(7):1315-1325. doi: 10.1136/gutjnl-2020-323476. Epub 2021 Aug 30. PMID 34462336